CLINICAL TRIAL: NCT05710653
Title: Physiological Response to a Training and Detraining Period in Vascular Parameters of Cardiometabolic Risk Factors Subjects: Optimizing Post-exercise Strategies to Maintain Health Benefits in Chilean Adults
Brief Title: Inter-individual Physiological Response to a Training and Detraining Period in Cardiometabolic Risk Factors Subjects
Acronym: VASCU-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristian Alvarez (Other)
Responsible Party: Sponsor-Investigator, Cristian Alvarez, Associate Professor, Universidad Nacional Andres Bello
Organization: Universidad Nacional Andres Bello (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAB-FCR-KINE2023A
Record Dates: First submitted 2023-01-20; First posted 2023-02-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Vascular Disease, Peripheral; Physical Inactivity; Arterial Hypertension; Endothelial Dysfunction
Keywords: Endothelial dysfunction; Exercise training; High-intensity interval training; Body composition; Exercise test; Obesity; Adults; Resistance training; Concurrent training
MeSH Terms: conditions — Peripheral Vascular Diseases; Sedentary Behavior; Hypertension; Obesity

STUDY DESIGN:
Intervention Model Description: We will compare three different exercise training experimental groups categories, such as; an arterial hypertension group (HTN), an elevated blood pressure (Ele), and a last normotensive (NT) experimental group in their physiological adaptations versus other three control groups of HTN, Ele, and NT control peers, after 3 months of training, and other 3 months od detraining y several health-related outcomes.
Who Masked: Participant, Investigator
Masking Description: According to availability and the feasibility of the enrolment's requirements, patients will be allocated to an arterial hypertension group (HTN), an elevated blood pressure (Ele), and a last normotensive (NT) experimental group, and thus randomly allocated to an experimental (HTNex, Eleex, NTex) or control group (HTNcg, Elecg, NTcg) in where subjetcs will not do HIIT exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HTNex (Experimental): The participants will adhere to 12 weeks of exercise training, three times a week.
  Interventions: Behavioral: Exercise training intervention
- HTNcg (No Intervention): These participants will maintain their normal lifestyle without intervention.
- ELEex (Experimental): The participants will adhere to 12 weeks of exercise training, three times a week.
  Interventions: Behavioral: Exercise training intervention
- ELEcg (No Intervention): These participants will maintain their normal lifestyle without intervention.
- NTex (Control Group-exercise) (Experimental): The participants will adhere to 12 weeks of exercise training, three times a week.
  Interventions: Behavioral: Exercise training intervention
- NTcg (Control Group-no exercise) (No Intervention): These participants will maintain their normal lifestyle without intervention.

INTERVENTIONS:
Behavioral: Exercise training intervention — The intervention will consist in adhering to high-intensity interval training and/or resistance training three times a week
  Other Names: Physical therapy intervention
  Arms: ELEex; HTNex; NTex (Control Group-exercise)

SUMMARY:
Background: Although exercise training is a well described therapy for some cardiometabolic diseases such as obesity, type 2 diabetes, arterial hypertension, and metabolic syndrome, there is scarcity of knowledge about the post-exercise period term as 'detraining' where usually all physiological adaptations as cardiovascular and metabolic benefits are lost due to physical inactivity. Likewise, as some exercise training modalities as high-intensity interval training improve vascular parameters including endothelial dysfunction parameters as flow-mediated dilation (FMD%), and carotid-intima media thickness (c-IMT) during the 'training' period, there is little knowledge about how many 'volume' or 'intensity' of exercise training or physical activity per week is needed to maintain the exercise training benefits in populations with cardiometabolic risk factors such as those patients with arterial hypertension. This information will be of great interest for both improving and maintaining the vascular profile and health of Chilean adults with risk factors and to maintain a better vascular profile. Objective: To study the beneficial adaptations from the 'training' and 'detraining' period of exercise training on functional and structural vascular parameters in healthy and cardiometabolic risk factors adult subjects to improve the health profile. Methods: The investigators will conduct an experimental design of 5 groups of exercise training in healthy (controls) and hypertensive (HTN) patients (≥140 mmHg), with overweight/or obesity, men and women, with BMI ≥25 and ≤35 kg/m2, aged ≥18y, physically inactive (<150 min/week of low/moderate PA/week, or <75 min/week of vigorous PA) in the last 6 months will be invited for participating. The groups will be as follows; Group (HTNex will be compared with Group HTNcg). Group (ELEex will be compared with Group ELEcg). Group (NTex will be compared with Group NTcg). Each group will be compared in their physiological vascular adaptations before and after exercise training such as HIIT, and after 3 months of a detraining period. Results (hypothesis): The investigators hypothesized that the maintenance of vascular outcomes after the 'detraining' period is intensity-dependent in adults with HTN that participated of an exercise intervention.

DETAILED DESCRIPTION:
Endothelial dysfunction (EDys) is characterized as a phenotypic alteration in the endothelium of the arteries, characterized by prothrombotic, pro-inflammatory, an imbalance between the actions of vasodilators and vasoconstrictors, and small resistance vessels. Functionally, the endothelium acquires a proinflammatory state, with prothrombic properties, and is commonly associated with cardiovascular diseases, such as arterial hypertension (HTN, i.e., higher SBP, DBP], coronary artery disease, chronic heart failure, peripheral artery disease, atherosclerosis, type 2 diabetes mellitus (T2DM), and chronic renal failure. Clinically, a decrease of 0.62% in the endothelial function, measured by flow-mediated dilation (FMD%), is associated with an increase of +20 mmHg in systolic blood pressure (SBP). Functionally, EDys is expressed by FMD%, pulse wave velocity (PWV), or the aortic augmentation index (AIx) of the brachial artery, and Structurally EDys is expressed by the carotid-intima media thickness (c-IMT) among others. Methodologically, both FMD% and c-IMT outcomes can be assessed by a) a non-invasive ultrasound, and b) by other more invasive technics.

Part of the mechanism that explains the reduced vasodilator capacity in EDys includes decreased nitric oxide (NO) production, increased oxidative stress (ROS), and a decrease in the production of hyperpolarizing factors. At the molecular level, the up-regulation of adhesion molecules, generation of macrophage chemoattractant peptide-1, and the production of plasminogen activator inhibitor-1 participate also in the inflammatory response related to the prothrombic state in EDys. Other molecular linked mechanisms include that angiotensin II and endothelin-1, hypercholesterolemia, altered insulin signaling, and hyperglycemia can contribute to EDys. Thus, EDys is a preliminary event before atherosclerosis, increasing plaque accumulation, involving molecular pathophysiological events, but also 'functional' and 'structural' detectable damage, that are highly linked with cardiovascular disease (CVD).

In this sense, the 'elevated' BP, clinically known as prehypertension (preHTN), and the HTN itself, represent an enormous public health issue, considering their high correlation with stroke, coronary heart disease, heart failure, and above to Chile, where there is accelerated aging of the population, where HTN is more common in older adults. The adult population with HTN have several other co-morbidities such as overweight/obesity (~40%), T2DM, and dyslipidemia (i.e. increased low-density lipids [LDL-c], decreased high-density lipids [HDL-c], or increased triglycerides), but are transversely physically inactive ~40% (i.e., to do not adhere to national and international physical activity/exercise training recommendations of at least 150 min/of physical activity/exercise training per week by the WHO guidelines).

Exercise training (ExT), a particular monitored modality of physical activity, can work by previous knowledge, as a 'therapy' for decreasing BP in HTN patients and in those with EDys. ExT is a planned, regulated, and guided physical activity modality, where participants can obtain benefits according to a dose applied (i.e., intensity, volume, frequency per week, density) and the profile (i.e., healthy, or seek with cardiometabolic diseases as HTN, dyslipidemia, T2DM, or others, increase fitness performance, but at the same time improve vascular and health markers such as FMD%, c-IMT, SBP/DBP, or MAP in HTN. ExT can include endurance training (ET), consisting of continuum exercise usually practice at low to 'moderate' intensity (walking/run/cycling/rowing, etc.), resistance training (RT), involving loads and external weights (dumbells, exercise machines with loads) with high impact on muscle and bone mass, but also with cardiovascular benefits as decreasing BP, and the last studied high-intensity interval training (HIIT) modality, which is a low-volume of briefs high-intensity intervals (usually cycling, rowing, or running) interspersed with recovery rest periods, and that show a time-efficient cardiometabolic health. All these three ExT modes have been shown to improve functionally, and structurally the EDys, to reduce BP, and improve several anthropometric, body composition, cardiovascular, metabolic, and physical fitness parameters in HTN patients, being this recently corroborated by the American Colleague of Sports Medicine.

Exercise training in Endothelial dysfunction: A relevant meta-analysis from Higashi et al. revealed that moderate-intensity of ET, increases the nitric oxide availability, promoting improvements in EDys markers in healthy subjects. A Long-term ET promote also regular endothelium-dependent vasodilation, and these physiological stimuli have been associated with lower blood pressure levels in HTN individuals. A very recently published article from Pedralli et al., where after 8-weeks of three different Ext modalities as ET, RT, and CT the authors showed a significant improvement in both BP and EDys markers in HTN patients. However, the relevance of these findings contain several scientific and methodological concerns to be considered and generalized such as a) there were no included the time-efficient exercise modality of HIIT, b) the investigators only reported FMD%, but not other of relevance to the endothelial function as c-IMT, c) there were no different frequencies groups of ExT/week, d) RT group worked at intensities ≥60% until 80% of the maximum strength in patients, the baseline PA level was reported by questionnaires rather than objectively measure PA using accelerometers devices, e) there was no diet control hour before the BP and EDys measurements, and more importantly, there was no control group and included both PreHTN, and HTN participants, among others (reported only results in 'mean', but not inter-individual response to know responders (Rs) and non-responders (NRs) to ExT modes. Additionally, and as a major concern, although there are some evidence that show significant improvements of vascular parameters from exercise training such as FMD% and c-IMT during the exercise-intervention periods, there is no evidence about how to maintain these physiological vascular benefits during 'detraining', where there is scarcity of studies with evidence about potential loss of these vascular adaptations, nor proposals of other minimum exercise-dose to maintain these vascular adaptations during the post-exercise cessation period.

Acute and long-term exercise training effects in BP and EDys markers: A single session of endurance training (ET) reduces resting blood pressure 5-7 mmHg among HTN patients, and this effect is sustained for up to 24h. This phenomenon is termed post-exercise hypotension effect. Ciolac et al. showed that 40 minutes of ET at 60% of the heart rate reserve, decreased SBP, and DBP day, and night, by using Holter monitors. Interestingly, the authors showed that there was an increase in the sample of HTN patients who showed normal daytime SBP (68% vs. 82), and nighttime diastolic blood pressure (56% vs. 72%). In HTN patients, after 60 minutes of ET (45 min, at 70% maximum oxygen consumption [VO2max]), Taylor-Tolbert et al. reduced SBP -7.4, and DBP -3.6 mmHg, maintaining up to 24h the PEHE. After an acute session of 60 minutes of ET, other authors had reported decreases in SBP -9.9 and DBP -6.2 mmHg in healthy Chilean adults. Cade et al. in 1984 reported that ET normalized BP, and decreased medications dosage in HTN patients after 12-weeks of training by decreasing SBP ~22, and DBP ~18 mmHg. However, after four decades of science and technological advances, there is wide evidence from different ExT modalities as ET, HIIT, or RT, in favor of normalizing (functionally) BP in HTN patients. Olea et al. have shown recently that after 24 sessions of HIT ExT, there was a reduction from 145 to 118 mmHg SBP in the HTN group, where the healthy normotensive group does not elicit changes. Interestingly, the authors reported a reduction of -3.9 kg of body fat, and from the 100% of the HTN sample (n=22), at the final of the ExT program, there was a 73% of patients that normalized (i.e., in the normotensive state) their SBP. Chen et al. reported that HTN patients decreased SBP -15, and DBP -4 mmHg after 12 months of 4-courses of sports. Previously, at long-term ExT on BP changes, our team have reported that long-term exercise training (≥4-weeks of regular exercise) in HTN patients decrease SBP -20, and DBP -9 mmHg BP after concurrent training (CT) of combining both HIT plus RT), decreasing SBP from 143 to 126 mmHg, and DBP from 83 to 71 mmHg in HTN patients. Other investigators have shown that 16-weeks of HIIT in PreHTN patients decrease SBP -8, DBP -5.8 mmHg, and healthy normotensive do not elicit changes. Interesting in this study, PreHTN patients decreased also -3.3 kg weight, -3 cm waist circumference, -5.8% body fat, -13.9 mg/dL triglycerides, increase +5.0 mg/dL HDL-c, increase +3 kg muscle strength in lower limbs, and improved their walking capacity by decreasing time in the 2 km walking test -3.1 min. After 12-weeks of ExT, other investigators reported significant decreases in PreHTN patients at SBP from RT -4 and HIT -6 mmHg, and in DBP -3 mmHg in HIT, wherein both ExT modalities reported significant improvements in obesity and physical fitness outcomes. However, after 20-weeks of ExT using CT (ET plus RT), HTN, and PreHTN patients can change their baseline diagnosis to another better stage, such as from HTN to PreHTN, or from PreHTN to normotension. These relevant and significant changes were accomplished by significant decreases in obesity, metabolic, and physical fitness markers. However, it was also reported that there was a wide IVET, where around ~30%, 50%, and 20% of patients in the CT exercise group showed no changes for improving body composition, blood pressure, and lipid profile, being named as nonresponders. Thus it is imperative to study more the ExT effects, such as HIIT and their physiological adaptations on EDys markers, and BP response in subjects with cardiometabolic risk factors such as those adults with preHTN, or HTN, but above the study of these parameters after a 'detraining' period and explore potential exercise dose to maintain the beneficial vascular adaptations and thus to protect the vascular system and overall health.

SARS Cov-2, Co-Morbidities and Exercise Training: The SARS Cov-2 viruses (COVID-19) have globally damage the overall physical and mental health in all the worldwide population. Unfortunately, although there are some asymptomatic subjects to the viruses, the main part of the death attributable to the COVID-19 virus are those with major co-morbidities such as population with obesity, HTN, cardiometabolic diseases and other with major respiratory diseases. Unfortunately, COVID-19 pandemic state have included a high physical inactivity situation that exacerbate the sedentary state and promote more impairment in blood pressure, and vasculature. Particularly, EDys is impaired in COVID-19, where the impairment of endothelial function have been related with more mortality risk in adults.

RESEARCH PROBLEM: Although there is relevant information about the ExT and their effects and mechanisms on EDys markers improvements such as at FMD% and c-IMT, there is little information regarding how long ExT in terms of 'volume' and 'intensity' can be able to maintain these ExT improvements after exercise cessation in a 'detraining' period testing a 'moderate', or a 'low' exercise dose of 'high' and 'low' exercise-intensity. This information could be useful for a decision to several ExT public health programs to the population with cardiometabolic risk factors for CVD, as well as to improve future more complex studies for predicting exercise response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, or subjects with elevated blood pressure (ELE) or arterial hypertension (HTN)
* ELE and/or HTN controlled or not controlled with pharmacotherapy
* With hyperglycemia, type 2 diabetes mellitus (T2DM) controlled or not controlled with pharmacotherapy
* Living in urban areas of the Concepción or Talcahuano cities
* Demonstrable ability to adhere to the exercise training programs
* To sign the written informed consent for participating in the study

Exclusion Criteria:

* Altered ECG
* Uncontrolled HTN (≥160 mmHg SBP, or DBP >95 mmHg)
* Morbid obesity (≥35-40 kg/m2)
* Type 1 diabetes mellitus
* Cardiovascular disease (i.e., coronary artery disease)
* T2DM complications such as varicose ulcer in the foot, legs, or any history of the wound, nephropathies, muscle-skeletal disorders (i.e., osteoarthrosis) that could limit exercise participation, and adaptations, where ExT can be not recommended.
* Subjects under pharmacotherapy that can influence body composition such as weight- loss treatment, as well as those who are enrolled in ExT programs recently (last 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation in (cm) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in flow-mediated dilation in the brachial artery registered by a linear transducer using images from a Doppler ultrasound
Pulse wave velocity in (m/s) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in pulse wave velocity in the brachial artery registered by an oscillometric cuff in the brachial artery
Carotid intima media thickness in (cm) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Carotid intima media thickness in common carotid artery registered by a linear transducer using images from a Doppler ultrasound

SECONDARY OUTCOMES:
Body mass in (kg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in body mass registered by a digital scale in kilograms
Height | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in height registered by a stadiometer in centimeters
Body mass index in (kg/m2) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in body mass index registered by from the calculation of the weight plus the height dividev by the suare of the height
Body fat in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in body fat percentage registered by from a digital bio-impedanciometer equipment
Skeletal muscle mass in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in skeletal muscle mass in percentage registered by from a digital bio-impedanciometer equipment
Resting metbolic rate in (kcal) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in resting metabolic rate obtained in kcalories from a digital bio-impedanciometer equipment
Body age in (years) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in body age estimated from a digital bio-impedanciometer equipment
Waist circumference in (cm) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in waist circumference obtained from a measuring tape in centimeters
Systolic blood pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position
Diastolic blood pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position
Mean arterial pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in mean arterial pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position, particularly from the data systolic and diastolic blood pressure obtained from this equipment
Pulse pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in pulse pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position, particularly from the data systolic and diastolic blood pressure obtained from this equipment
Heart rate at rest in (beats/min) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in heart rate at rest obtained from a digital watch cardiometer in beats/min
Systolic blood pressure of the ankle in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic blood pressure of the ankle in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Partial oxygen saturation in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Partial oxygen saturation in (%) obtained from a digital saturometer from the index finger in seated position
Total chlesterol in (mg/dL) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in total cholesterol in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Fasting glucose in (mg/dL) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in fasting glucose in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Triglycerides in (mg/dL) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in triglycerides in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Augmentation index in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Augmentation index in (%) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Ankle-Brachial Index in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Ankle-Brachial Index in (%) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic Systolic blood pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Aortic Systolic blood pressure in (mmHg) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic pulse pressure in (mmHg) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Aortic pulse pressure in (mmHg) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic augmentation index in (%) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Aortic augmentation index in (%) obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Ejection duration in (m/s) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Ejection duration in (m/s) obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic reflection area | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Diastolic reflection area obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Systolic area index | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Systolic area index obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic area index | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Diastolic area index obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Return time of the aortic pulse wave | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in Return time of the aortic pulse wave measured in the brachial artery obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Arterial age | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Change in arterial age estimated from a digital cuff Arteriograph equipment measured from the brachial artery
Heart rate during exercise in (beats/min) | Baseline, 6 weeks, 12 weeks after exercise training intervention, and after 6 weeks, and 12 weeks follow-up
  Heart rate measured using a cardiometer watch equipment at different power output intensities using an cycle ergometer equipment

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Araneda, PhD, Study Chair — Universidad Andres Bello
Locations (1):
- Universidad Andres Bello, Talcahuano, Chile

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT05710653/Prot_SAP_000.pdf